CLINICAL TRIAL: NCT05880888
Title: Investigating the Clinical Impact of a Novel Adipose Allograft Matrix on Knee Fat Pad Impingement Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Baria, Associate Professor of Physical Medicine and Rehabilitation, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023H0043
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Fat Pad Syndrome
Keywords: Fat Pad Impingement; Adipose Allograft Matrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Renuva Injection (Experimental): Each subject will receive a single injection of up to 3ccs of Renuva into their diseased fat pad.
  Interventions: Biological: Renuva

INTERVENTIONS:
Biological: Renuva — Renuva® (MTF Biologics) is an injectable decellularized allograft adipose matrix (AAM) used to increase volume in adipose tissue.

SUMMARY:
This study is to assess the effect of Renuva® on fat pad regeneration in patients with Fat pad Impingement

DETAILED DESCRIPTION:
The fat pad of the knee works to stabilize the patella and releases cytokines, growth factors, and stem cells. These cytokines, growth factors, and stem cells exhibit anti-inflammatory, anabolic effects that can be recruited to heal the articular tissues of the knee and ameliorate their catabolic effects during osteoarthritis (OA).

The majority of the current treatments for fat pad impingement (FPI) and its sequelae are primarily symptom-modifying, and structure-modifying therapies both at the joint and peri-articular structures levels cannot be overemphasized.

Renuva® (MTF Biologics) is a Food and Drug Administration approved, off-the-shelf, injectable decellularized allograft adipose matrix (AAM) used to increase volume in adipose tissue. Once injected, native cell populations infiltrate the AAM, and over time, the AAM remodels into native tissue and stimulates both adipogenesis and angiogenesis within the tissue.

Our specific aim is to assess the effect of Renuva® on fat pad regeneration in patients with FPI. The investigators hypothesize that injection of Renuva® into a diseased fat pad of the knee increase the volume of the fat pad and reduce any hemorrhage, edema or fibrosis present, when pre-to post-treatment images are compared.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age
* Fat pad impingement
* Knee MRI taken before study enrollment
* Working knowledge of English language (to be able to complete all outcome scores)
* Ability to attend all follow-up appointments.
* Able to undergo MRI

Exclusion Criteria:

* Medical condition that may impact outcomes of procedure including:

  * Systemic inflammatory disorders that impact the joints like rheumatoid arthritis, lupus, etc
  * Undergoing current cancer treatment (other than non-melanoma skin malignancies)
* Gout, Pseudogout (including radiographic evidence of chondrocalcinosis)
* History of infection or current infection at the affected joint
* Smoking (Former smokers< 1 year from quit date)
* Significant allergies manifested by a history of anaphylaxis or severe allergen sensitivity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-04-22 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Knee MRI measurements of fat pad thickness (mm) | 6 Months
  Knee MRI will be taken at 6 months post injection to compare the fat pad thickness (mm) to the MRI taken prior to the injection of Renuva.
Knee MRI measurements of fat pad surface area (mm2) | 6 Months
  Knee MRI will be taken at 6 months post injection to compare the fat pad surface area (mm2) to the MRI taken prior to the injection of Renuva.
Knee MRI measurements of fat pad volume (mm3) | 6 Months
  Knee MRI will be taken at 6 months post injection to compare the fat pad volume to the MRI taken prior to the injection of Renuva.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) Pain patient reported outcome questionnaire | 6 Months
  KOOS Pain evaluates short-term and long-term pain in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee pain.
Knee injury and Osteoarthritis Outcome Score (KOOS) Symptoms patient reported outcome | Baseline, 1 month, 3 month and 6 month
  KOOS symptoms evaluates short-term and long-term symptoms in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee symptoms.
Knee injury and Osteoarthritis Outcome Score (KOOS) Function in daily living (ADL) patient reported outcome | Baseline, 1 month, 3 month and 6 month
  KOOS ADL evaluates short-term and long-term function in daily living in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee related issues in regards to daily living activity.
Knee injury and Osteoarthritis Outcome Score (KOOS) Function in Sport and Recreation (Sport/Rec) patient reported outcome | Baseline, 1 month, 3 month and 6 month
  KOOS Sport/Rec evaluates short-term and long-term function in sports and recreation in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee related issues in regards to sports or recreation activity.
Knee injury and Osteoarthritis Outcome Score (KOOS) knee related quality of life (QOL) patient reported outcome | Baseline, 1 month, 3 month and 6 month
  KOOS QOL evaluates short-term and long-term knee quality of life in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee related issues in regards to quality of life.
Knee injury and Osteoarthritis Outcome Score (KOOS) Pain patient reported outcome | Baseline, 1 month, 3 month and 6 month
  KOOS Pain evaluates short-term and long-term pain in subjects with knee injury and osteoarthritis. Scores range from 0-100 where 100 represents no knee pain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baria, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Jameson Crane Sports Medicine Institute, Columbus, Ohio
  - Ohio State Outpatient Lewis Center, Lewis Center, Ohio

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared